CLINICAL TRIAL: NCT00644059
Title: A Phase III, Randomized, Observer-blind, Controlled, Multi-center Clinical Trial to Evaluate the Efficacy, Safety and Immunogenicity of One and Two Intramuscular Doses of Influenza Vaccine Versus Control Vaccines in Healthy Subject Aged 6 to <72 Months
Brief Title: Study to Evaluate the Efficacy, Safety and Immunogenicity of Influenza Vaccine in Healthy Subjects (Aged 6 to <72 Months) Versus Control Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P5; Eudract number 2007-003786-41; NCT01015885 (obsolete NCT alias)
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Influenza, Human
Keywords: Influenza; vaccine; children
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; serogroup C meningococcal conjugate vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TIV-adj (Experimental): Adjuvanted trivalent inactivated subunit influenza vaccine
  Interventions: Biological: Adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control (Active Comparator): Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
  Interventions: Biological: Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-flu Control (Sham Comparator): Novartis meningococcal C conjugate vaccine or tick-borne encephalitis vaccine
  Interventions: Biological: Meningococcal C conjugate vaccine or tick-borne encephalitis vaccine

INTERVENTIONS:
Biological: Adjuvanted trivalent inactivated subunit influenza vaccine — Either two intramuscular (IM) injections of half dose or one IM injection of full dose, depending on age of subject, were administered in the deltoid muscle preferably of the non-dominant arm.
  Other Names: Fluad
  Arms: TIV-adj
Biological: Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine — For both vaccines, either two intramuscular (IM) injections of half dose or one IM injection of full dose, depending on age of subject, were administered in the deltoid muscle preferably of the non-dominant arm.
  Other Names: 1) Agrippal; 2) Influsplit SSW
  Arms: Flu-control
Biological: Meningococcal C conjugate vaccine or tick-borne encephalitis vaccine — 1. Meningococcal vaccine: two IM injections
  2. Tick-borne encephalitis vaccine: two IM injections
  Other Names: 1. Menjugate; 2. Encepur Children
  Arms: Non-flu Control

SUMMARY:
This study will evaluate the efficacy, safety and immunogenicity of one or two 0.25 mL or 0.5 mL intramuscular injections of an adjuvanted influenza vaccine compared with non-influenza and non-adjuvanted influenza control vaccines in subjects 6 to <72 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Children whose parents/legal guardians have given written informed consent prior to study entry: a) aged 6 to <72 months (Part I and II of the study; influenza seasons 2007/2008 and 2008/2009) b) aged 6 to <36 months (Part III of the study; influenza season 2009/2010)
* In good health as determined by: a) medical history, b) physical examination, c) clinical judgment of the investigator

Exclusion criteria:

* Administration of licensed vaccines (including H1N1sw vaccines) within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study. Routine vaccines, according to local recommendations, or any other vaccines not foreseen in the protocol could be given after the active trial phase (i.e., 21 days after last vaccination) has been concluded.
* Receipt of another investigational vaccine or any investigational agent within 30 days prior to enrollment in the study or before completion of the safety follow-up period in another study, whichever is longer, and participation in another clinical trial during the present study.
* Experience of a severe acute infectious disease in the month prior to study start or experience of a mild acute infection disease in the week prior the study start (untreated common cold is acceptable). The severity of the infectious disease occurred will be based on the investigator's judgment.
* Any severe acute respiratory disease and infection requiring systemic antibiotic or antiviral therapy ongoing or resolved within 2 days prior to study start.
* Experience an axillary temperature equal to or greater than 37.8°C (rectal temperature equal to or greater than 38.3°C) within the 2 days before enrollment.
* Any serious disease in the opinion of the investigator including, for example: a) cancer, b) autoimmune disease (including rheumatoid arthritis under immunosuppressive therapy), c) insulin dependent diabetes mellitus, d) chronic pulmonary disease, asthma under inhalative therapy only is acceptable, e) acute or progressive hepatic disease, f) acute or progressive renal disease.
* Known or suspected impairment/alteration of immune function, for example, resulting from: a) receipt of immunosuppressive therapy (corticosteroid -except topical or inhaled steroids- or cancer chemotherapy), b) receipt of immunostimulants, c) receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 90 days and for the full length of the study, d) high risk for developing an immunocompromising disease (suspected or known HIV infection or HIV-related disease).
* Bleeding diathesis.
* History of hypersensitivity to any component of the study medication or chemically related substances.
* History of any anaphylaxis, serious vaccine reactions, or allergy to eggs, egg products or any other vaccine component.
* Laboratory confirmed influenza disease.
* History of neurological disorder or seizures (febrile seizures allowed).
* Received any influenza vaccine.
* Major surgery planned during the study period.
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives, e.g., planned travel or relocation of residence that would interfere with completion of study.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4902 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vacccines and Diagnostics, Study Director — Novartis
Locations (101):
- Finland (17):
  - East Vantaa Clinic, East Vaanta
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - Kotka Clinic, Kotka
  - Kuopio Vaccine Clinic, Kuopio
  - Kuopio Vaccine Research Clinic, Kuopio
  - Lahti vaccine research Clinic, Lahti
  - Oulu Vaccine Research Clini, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinajoki Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Clinic, Turku
  - Vantaa West Vaccine Research Clinic, Vantaa
  - West Vantaa Clinic, West Vantaa
- Germany (82):
  - Johannes Gutenberg-University, Mainz, Mainz
  - Praxis Dr med Thilo Heising, Aalen Wasseralfingen
  - Praxis Dr med Ursula Hornlein, Berlin
  - Praxis Dr med Thomas Richter, Berlin
  - Praxis Dipl med Andreas Muhmer, Berlin
  - Praxis Dr med Mechthild Vocks-Hauck, Berlin
  - Praxis Dr med Klaus-Peter Falkowski, Berlin
  - Praxis Dr med Eva Brand, Berlin
  - Praxis Dr med Dorothea Budde, Berlin
  - Praxis Dr. med. Cornelia Busse, Berlin
  - Praxis Dipl. med. F. Temmler / Dipl. med. D. Wenzel, Berlin
  - Praxis Dr med Petra van Stiphout, Berlin
  - Praxis Dr Luise Schroeter, Berlin
  - "Praxis Dr med Dietrich Lasius", Berlin
  - Praxis Dr. med. Petra Sandow, Berlin
  - Praxis Dr Norbert Meister, Bindlach
  - Praxis Dr med Thomas Tuschen, Binngen Rhein
  - Praxis Dr. Elmar Dietmair, Bobingen
  - Praxis Dr med Brigitta Becker, Bochum
  - Praxis Karl-Heinz Blattel, Braunfels
  - Praxis Dr. med. Roland Knecht, Bretten
  - Praxis Dr. med. Maria R. Holtorf, Brunsbüttel
  - Praxis Dr Klaus Helm, Detmold
  - Praxis Joseph Zakarian, Düsseldorf
  - Praxis Dr med Hans-Henning Peters, Eschwege
  - Praxis Dr. med. Dirk Straub, Essen
  - Praxis Dr med Rainer Haase, Flensburg
  - Praxis Dr. med. Per Gildberg, Flensburg
  - Peaxis Dr H Outzen jun, Flensburg
  - Praxis Dr Lothar MaurerJun, Frankenthal
  - Praxis Dr med Walter Otto, Fulda
  - Praxis Dr med Hans-Joachim Buttner, Gau-Odernheim
  - Praxis Dr med Christian Kayser, Gehrden
  - Praxis Ute Jessat, Glücksburg
  - Praxis Dr. med. Dubravka Pock-Lutz, Grevenbroich
  - Praxis Dr. med. Malte Klarczyk, Hamburg
  - Praxid Dr. med. Karl-Heinrich Hansen, Hamburg
  - Praxis Dr Anna Halat, Hamburg
  - Praxis Dr med Bernard Nast, Hamburg
  - Praxis Dr med Jurgen Schwalbe, Hamelin
  - Praxis Dr med Hans-Heinrich Rohe, Hille
  - Praxis Dr Marlies Bolich, Jena
  - Praxis Peter Bosch, Karlsruhe-Oberreut
  - Praxis Dr Peter Andoko Soemantri, Kleve-Materborn
  - Praxis Dr. Michael Muehlschlegel, Lauffen am Neckar
  - Praxis Dr Sibylle Hetzinger, Lobenstein
  - Praxis Dipl med Dagmar Manegold-Randel, Löhne
  - Praxis Dr. Renate Lang, Ludwigsburg
  - Praxis Dr med Julika Kelber, Lüneburg
  - Praxis Uwe Jakob, Mainz
  - Praxis Dr med Falko Panzer, Mannheim
  - Praxis Dr med Volker Tempel, Marbach A. N.
  - Praxis Dr. med. Herbert Kollaschinski, Marktredwitz
  - Praxis Dr med Matthias Donner, Mönchengladbach
  - Praxis Ralph Koellges, Mönchengladbach
  - Praxis Dr med Philip Fellner von Feldegg, Munster / NRW
  - Praxis Dr. med. Janina Joiko, München
  - "Praxis Prof Dr med Stefan Walter Eber", München
  - Praxis Dr med Peter Dietl, München
  - Praxis Dipl Med Ute Macholdt, Neuhaus am Rennweg
  - Praxis Dr Rossius, Neumünster
  - Praxis Dr Sabine Maruschke, Neumünster
  - Praxis Drs J und K Kandzora, Neumünster
  - Praxis Dr. med. S. Mohns-Petersen, Niebüll
  - Praxis Dr med Hartmut Scheele, Niedernhausen
  - Praxis Dr med Stefan Noll, Porta Westfalica
  - Praxis Zlatka Zochev Donkov, Rendsburg
  - Praxis Thomas Morandini, Schönenberg
  - Praxis Dr med Michael Vomstein, Schwäbisch Hall
  - "Praxis Dr med Gunther Knapp", Schwieberdingen
  - Praxis Dr med Ulrich Soergel, Stadthagen
  - Praxis Dr Ulrich Pfletschinger, Stuttgart
  - Praxis Dr. med Manfred Heitz, Stuttgart
  - Praxis Dr. med Heidi B. John-Wagenmann, Stuttgart
  - Praxis Dr. med. Rolf Ebert, Tauberbischofsheim
  - Praxis Dr med Karl-Eugen Mai, Tettnang
  - Praxis Dr med Klaus Kindler, Trier
  - Praxis Dr med Ralph Maier, Tuttlingen
  - Praxis Dr med Ulrich Umpfenbach, Viersen
  - Praxis Dr med Volker Kemmerich, Weinstadt
  - Praxis Dr Per Bergmann, Winsen
  - Praxis Dr med Steffi Bulst, Wurzen
- Italy (2):
  - Fondazione IRCCS Policlinico Mangiagalli e Regina Elena, Milan
  - Ospedale Maggiore della Carita, Novara

REFERENCES:
- [Result] Vesikari T, Knuf M, Wutzler P, Karvonen A, Kieninger-Baum D, Schmitt HJ, Baehner F, Borkowski A, Tsai TF, Clemens R. Oil-in-water emulsion adjuvant with influenza vaccine in young children. N Engl J Med. 2011 Oct 13;365(15):1406-16. doi: 10.1056/NEJMoa1010331. PMID 21995388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled as follows:
  In season 2007/08: 28 active sites in Germany (Excluding Site 023); In season 2008/09: 83 active sites+ 1 coordinating site in Germany, 15 sites in Finland; In season 2009/10: 15 sites in Finland, 2 sites in Italy
Pre-assignment Details: All subjects enrolled were included in the trial. The data entered is for the overall study.
Groups:
- TIV-adj: Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control: Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-flu Control: Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of Tick-borne encephalitis (TBE) vaccine
Period: Overall Study
Arm/Group | TIV-adj | Flu-control | Non-flu Control
Started | 2019 | 1849 | 1034
Completed | 1895 | 1726 | 969
Not Completed | 124 | 123 | 65
Not completed — Lost to Follow-up | 37 | 34 | 16
Not completed — Withdrawal by Subject | 52 | 60 | 30
Not completed — Adverse Event | 8 | 5 | 1
Not completed — Inappropriate Enrollment | 1 | 3 | 0
Not completed — Protocol Deviation/violation | 20 | 19 | 15
Not completed — Unable to classify | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Non-flu Control: Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
- Total: Total of all reporting groups
Arm/Group | TIV-adj | Flu-control | Non-flu Control | Total
Number analyzed (Participants) | 2019 | 1849 | 1034 | 4902
Age, Continuous [Mean (Standard Deviation); unit: Months] | 31.9 (19.8) | 32.6 (20.1) | 32.2 (19.8) | 32.2 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 962 | 903 | 484 | 2349
  Male | 1057 | 946 | 550 | 2553

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects (Unprimed) 6 to <36 Months Age With Local and Systemic Reactions After Any Vaccination for All Seasons, Comparison of Adjuvanted Trivalent Influenza Vaccine (aTIV) and Flu Vaccine Control.
Description: Safety was assessed in terms of number of subjects experiencing each of the local and systemic reactions within 7-days after any vaccination for all seasons, comparison of adjuvanted Trivalent influenza vaccine (aTIV) and flu vaccine control.
Time Frame: 7 days post-vaccination
Population: The analysis was done on Safety set - All subjects in the exposed population who provided post-baseline safety data.
Measure: Number; unit: Number of subjects
Groups:
- TIV-adj (6 to <36 Months): Subjects aged 6 to <36 months received 0.25 mL of each injection of Adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control (6 to <36 Months): Subjects aged 6 to <36 months received 0.25 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
Arm/Group | TIV-adj (6 to <36 Months) | Flu-control (6 to <36 Months)
Number analyzed (Participants) | 1178 | 1068
Number of subjects
  Any Local | 625 | 481
  Injection Site Ecchymosis | 147 | 103
  Injection Site Erythema | 423 | 322
  Injection Site Induration | 214 | 131
  Swelling | 123 | 89
  Tender. at inj.site | 330 | 246
  Any Systemic | 785 | 694
  Change in eat. hab. | 325 | 261
  Sleepiness | 380 | 312
  Unusual crying | 386 | 345
  Irritability | 387 | 353
  Vomiting | 131 | 118
  Diarrhea | 258 | 211
  Shivering | 77 | 69
  Any Other | 358 | 317
  Fever (38-38.9°C) (N=1177,1068) | 169 | 143
  Fever (39-39.9°C) (N=1177,1068) | 61 | 43
  Fever (>40.0°C) (N=1177,1068) | 3 | 3
  Analg.Antipyr.Used (N=1176,1068) | 358 | 317

2. Primary Outcome: Percentage of Subjects (Unprimed) Aged 6 to <36 Months With Virus-Confirmed Influenza, Comparison of aTIV and Non-flu Vaccine Control (Men C/TBE Vaccine)
Description: Virus-confirmed influenza illnesses were assessed and compared between the adjuvanted influenza vaccine (TIV-adj) and non-influenza vaccines (Non-flu control) in 6 to <36 month unprimed subjects for Absolute Efficacy. This primary endpoint is only for homologous strains.
Time Frame: 3 weeks after 2nd vaccination
Population: Analysis was done on Full Analysis Set (FAS) - All subjects in the enrolled set who received study vaccination and provided at least one evaluable serum sample both before and after baseline.
Measure: Number; unit: Percentage of subjects
Groups:
- TIV-adj (6 to <36 Months): Subjects aged 6 to < 36 months received 0.25 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Non-flu Control (6 to <36 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
Arm/Group | TIV-adj (6 to <36 Months) | Non-flu Control (6 to <36 Months)
Number analyzed (Participants) | 916 | 469
Percentage of subjects
  Season 2007/2008, Matched strain,N=187,97 | 0 | 0
  Season 2008/2009, Matched strain | 0.76 | 4.05
Statistical Analysis 1: Comparison: TIV-adj (6 to <36 Months) vs Non-flu Control (6 to <36 Months); Absolute vaccine efficacy (VE) was calculated as (1- the relative risk)100%. Relative Risk for virus-confirmed symptomatic influenza illness in the TIV-adj group vs. the non-flu control group. VE denotes the vaccine efficacy, i.e. 1-Itest/Inon-flu ctrl, where I stands for the population average incidence of influenza. Absolute efficacy of TIV-adj is at most 40% (i.e. the probability of an influenza in the test group relative to that in the non-flu vaccine group is at least 0.6); Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 81.36, 97.66% CI 2-sided [49.24 to 93.16]

3. Secondary Outcome: Number of Subjects (Unprimed) of 6 to <72 Months Age With Local and Systemic Reactions After Any Vaccination
Description: Safety was assessed as the number of subjects aged 6 to <72 months who reported solicited local or systemic adverse events after any vaccination with TIV-adj for all seasons.
Time Frame: 7 days post-vaccination
Population: The analysis was done on Safety set
Measure: Number; unit: Number of subjects
Groups:
- TIV-adj (36 to <72 Months): Subjects aged 36 to < 72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control (6 to <36 Months): Subjects aged 6 to < 36 months received 0.25 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Flu-control (36 to <72 Months): Subjects aged 36 to < 72 months received 0.5 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-Flu-control (6 to <36 Months); Non-Flu-control (36 to <72 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
Arm/Group | TIV-adj (6 to <36 Months) | TIV-adj (36 to <72 Months) | Flu-control (6 to <36 Months) | Flu-control (36 to <72 Months) | Non-Flu-control (6 to <36 Months) | Non-Flu-control (36 to <72 Months)
Number analyzed (Participants) | 1178 | 833 | 1068 | 778 | 607 | 422
Number of subjects
  Any Local | 625 | 569 | 481 | 466 | 315 | 232
  Inj. site ecchymosis(N=1178,833,1068,777,607,422) | 147 | 130 | 103 | 93 | 69 | 49
  Inj. site erythema(N=1178,833,1068,777,607,422) | 423 | 320 | 322 | 269 | 239 | 129
  Inj. site induration(N=1178,833,1068,777,607,422) | 214 | 168 | 131 | 152 | 153 | 80
  Inj. site swelling(N=1178,833,1068,777,607,422) | 123 | 155 | 89 | 128 | 82 | 55
  Inj. site tenderness(N=1178,0,1068,0,607,0) | 330 | 0 | 246 | 0 | 171 | 0
  Inj. site pain (N=0,833,0,777,0,422) | 0 | 477 | 0 | 360 | 0 | 180
  Any Systemic | 785 | 523 | 694 | 341 | 370 | 211
  Change in eat. hab.(N=1178,0,1068,0,607,0) | 325 | 0 | 261 | 0 | 162 | 0
  Sleepiness (N=1178,0,1068,0,607,0) | 380 | 0 | 312 | 0 | 186 | 0
  Unusual crying (N=1178,0,1068,0,607,0) | 386 | 0 | 345 | 0 | 175 | 0
  Irritability (N=1178,0,1068,0,607,0) | 387 | 0 | 353 | 0 | 187 | 0
  Vomiting (N=1178,0,1068,0,607,0) | 131 | 0 | 118 | 0 | 66 | 0
  Diarrhea (N=1178,0,1068,0,607,0) | 258 | 0 | 211 | 0 | 114 | 0
  Shivering (N=1178,0,1068,0,607,0) | 77 | 0 | 69 | 0 | 50 | 0
  Chills shivering (N=0,833,0,777,0,422) | 0 | 130 | 0 | 51 | 0 | 37
  Malaise (N=0,833,0,777,0,422) | 0 | 196 | 0 | 118 | 0 | 63
  Myalgia (N=0,833,0,777,0,422) | 0 | 183 | 0 | 100 | 0 | 66
  Arthralgia (N=0,833,0,777,0,422) | 0 | 82 | 0 | 37 | 0 | 27
  Headache (N=0,833,0,777,0,422) | 0 | 197 | 0 | 100 | 0 | 54
  Sweating (N=0,833,0,777,0,422) | 0 | 69 | 0 | 42 | 0 | 31
  Fatigue (N=0,833,0,777,0,422) | 0 | 337 | 0 | 222 | 0 | 123
  Any Other | 358 | 196 | 317 | 94 | 159 | 69
  Fever(38-38.9C)(N=1177,833,1068,775,607,421) | 169 | 133 | 143 | 55 | 62 | 37
  Fever(39-39.9C)(N=1177,833,1068,775,607,421) | 61 | 50 | 43 | 17 | 34 | 19
  Fever(≥40.0C)(N=1177,833,1068,775,607,421) | 3 | 1 | 3 | 2 | 2 | 1
  Analg.Antipyr.Used (N=1176,833,1068,777,607,422) | 358 | 196 | 317 | 94 | 159 | 69

4. Secondary Outcome: Number of Subjects (Unprimed) With Unsolicited Adverse Events Reported After Any Vaccination
Description: Number of subjects aged 6 to <36 months and in the overall age cohort (unprimed children aged 6 to <72 months) experiencing each of the unsolicited adverse events (AEs) throughout the study
Time Frame: Study day 1 to Study day 181
Population: The analysis was done on Safety set
Measure: Number; unit: Number of subjects
Groups:
- TIV-adj (6 to <72 Months ): Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control (6 to <72 Months): Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-Flu-control (6 to <72 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
Arm/Group | TIV-adj (6 to <36 Months) | Flu-control (6 to <36 Months) | Non-Flu-control (6 to <36 Months) | TIV-adj (6 to <72 Months ) | Flu-control (6 to <72 Months) | Non-Flu-control (6 to <72 Months)
Number analyzed (Participants) | 1177 | 1069 | 607 | 2012 | 1846 | 1029
Number of subjects
  Any AEs | 1045 | 938 | 530 | 1714 | 1566 | 867
  At least possibly related AEs | 152 | 124 | 90 | 262 | 203 | 137
  Serious AEs | 91 | 104 | 65 | 122 | 169 | 110
  At least possibly related SAEs | 1 | 1 | 3 | 2 | 2 | 3
  AEs leading to discontinuation | 6 | 9 | 1 | 9 | 10 | 1

5. Secondary Outcome: Percentage of Subjects (Unprimed) Aged 6 to <72 Months With Virus-Confirmed Influenza, Comparison of aTIV to Non-flu Vaccine Control and Flu-vaccine Control (Matched Strains)
Description: Virus-confirmed influenza illnesses were assessed and compared between the adjuvanted influenza vaccine (TIV-adj) and non-influenza vaccines (Non-flu control) in subjects aged 6 to <72 months (unprimed) for Absolute Efficacy.
  For Relative efficacy, the comparison was made between adjuvanted influenza vaccine (TIV-adj) and flu vaccine control.
Time Frame: 3 weeks after 2nd vaccination
Population: The analysis was done on Full Analysis Set
Measure: Number; unit: Percentage of subjects
Groups:
- TIV-adj (6 to < 36 Months): Subjects aged 6 to < 36 months received 0.25 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu Control (6 to < 36 Months): Subjects aged 6 to < 36 months received 0.25 mL of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- TIV-adj (36 to < 72 Months): Subjects aged 36 to < 72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Non-flu Control (36 to <72 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
- Flu Control (36 to < 72 Months): Subjects aged 36 to < 72 months received 0.5 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
Arm/Group | TIV-adj (6 to < 36 Months) | Non-flu Control (6 to <36 Months) | Flu Control (6 to < 36 Months) | TIV-adj (36 to < 72 Months) | Non-flu Control (36 to <72 Months) | Flu Control (36 to < 72 Months)
Number analyzed (Participants) | 916 | 469 | 902 | 698 | 360 | 706
Percentage of subjects
  Matched strain(Season2007/08)N=187,97,93,136,67,71 | 0 | 0 | 0 | 0 | 0 | 0
  Matched strain (Season2008/09) | 0.76 | 4.05 | 2.44 | 0.29 | 6.11 | 3.12
Statistical Analysis 1: Comparison: TIV-adj (6 to < 36 Months) vs Non-flu Control (6 to <36 Months); Absolute vaccine efficacy (VE) was calculated as (1- the relative risk)100%. Relative Risk for virus-confirmed symptomatic influenza illness in the TIV-adj group vs. the non-flu control group. VE denotes the vaccine efficacy, i.e. 1-Itest/Inon-flu ctrl, where I stands for the incidence of influenza. Absolute efficacy of TIV-adj is at most 40% (i.e. the probability of an influenza in the test group relative to that in the non-flu vaccine group is at least 0.6); Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 81.36, 95% CI 2-sided [49.24 to 93.16]
Statistical Analysis 2: Comparison: TIV-adj (36 to < 72 Months) vs Non-flu Control (36 to <72 Months); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 95.5, 95% CI 2-sided [80.92 to 98.94]
Statistical Analysis 3: Comparison: TIV-adj (6 to < 36 Months) vs Flu Control (6 to < 36 Months); Relative efficacy for TIV-adj was to be calculated as VE = (1-Itest/Ictrl)100%, where I is the incidence of influenza, i.e. percentage of subjects with virus-confirmed symptomatic influenza A or B illness, in the investigational agent (TIV-adj) group or in the flu vaccine control group; Test type: Superiority or Other; Mantel Haenszel; Vaccine Efficacy = 0.32, 95% CI 2-sided [0.13 to 0.73]
Statistical Analysis 4: Comparison: TIV-adj (36 to < 72 Months) vs Flu Control (36 to < 72 Months); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; Mantel Haenszel; Vaccine Efficacy = 0.09, 95% CI 2-sided [0.02 to 0.38]

6. Secondary Outcome: Percentage of Subjects (Unprimed) Aged 6 to <72 Months With Virus-Confirmed Influenza, Comparison of aTIV to Non-flu Vaccine Control and Flu Vaccine Control (Any Strains).
Description: Virus-confirmed influenza illnesses (regardless of antigenic match to those contained in the vaccine) were assessed and compared between the adjuvanted influenza vaccine (TIV-adj) and non-influenza vaccines (Non-flu control) in subjects aged 6 to <72 months (unprimed) for Absolute Efficacy.
  For Relative efficacy, the comparison was made between adjuvanted influenza vaccine (TIV-adj) and flu vaccine control.
Time Frame: 3 weeks after 2nd vaccination
Population: Analysis was done on Full Analysis Set
Measure: Number; unit: Percentage of subjects
Groups:
- Non-flu Control (6 to < 36 Months); Non-flu Control (36 to < 72 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
- Flu Control (6 to < 36 Months): Subjects aged 6 to < 36 months received 0.25 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
Arm/Group | TIV-adj (6 to < 36 Months) | Non-flu Control (6 to < 36 Months) | Flu Control (6 to < 36 Months) | TIV-adj (36 to <72 Months) | Non-flu Control (36 to < 72 Months) | Flu Control (36 to < 72 Months)
Number analyzed (Participants) | 916 | 469 | 902 | 698 | 360 | 706
Percentage of subjects
  Any Strain (Season 2007/08)N=187,97,93,136,67,71 | 0 | 2.06 | 0 | 0.74 | 2.99 | 0
  Any Strain (Season 2008/09) | 0.98 | 4.26 | 2.77 | 0.43 | 6.39 | 3.54
Statistical Analysis 1: Comparison: TIV-adj (6 to < 36 Months) vs Non-flu Control (6 to < 36 Months); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Poisson Regression Model; vaccine Efficacy = 79.18, 95% CI 2-sided [54.78 to 90.42]
Statistical Analysis 2: Comparison: TIV-adj (36 to <72 Months) vs Non-flu Control (36 to < 72 Months); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 92.1, 95% CI 2-sided [77.35 to 97.24]
Statistical Analysis 3: Comparison: TIV-adj (6 to < 36 Months) vs Flu Control (6 to < 36 Months); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 64.16, 95% CI 2-sided [23.21 to 83.28]
Statistical Analysis 4: Comparison: TIV-adj (36 to <72 Months) vs Flu Control (36 to < 72 Months); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; Poisson Regression Model; Vaccine Efficacy = 85.66, 95% CI 2-sided [58.95 to 94.99]

7. Secondary Outcome: Number of Subjects (Unprimed) With Influenza Like Illnesses (ILIs) in the 6 to <72 Months Age Cohort for Combined Seasons 2007/08 and 2008/09
Description: Virus-confirmed influenza illnesses were assessed and trivalent adjuvanted influenza vaccine (TIV-adj) was compared with Non-flu control vaccine and Flu-control vaccine in 6 to <72 month old subjects for Influenza like illnesses for seasons 2007/08 and 2008/09.
Time Frame: 3 weeks after 2nd vaccination
Population: Analysis was done on Full Analysis Set
Measure: Number; unit: Number of subjects
Arm/Group | TIV-adj | Flu-control | Non-flu Control
Number analyzed (Participants) | 1937 | 1772 | 993
Number of subjects
  Subjects with ILI | 425 | 436 | 253
  Outpatient visits | 290 | 293 | 174
  Inpatient visits | 20 | 26 | 19
  Outcome (Recovered) | 414 | 431 | 248
  Outcome (Alive with sequelae) | 5 | 2 | 2
  Outcome (Lost to follow-up) | 3 | 1 | 0
  Outcome (ILI persisting) | 3 | 1 | 3
  Outcome (Not available) | 0 | 1 | 0

8. Secondary Outcome: Number of Subjects With Influenza Like Illnesses (ILIs) in the 6 to <36 Months and in Overall Age Cohort (Unprimed Subjects Aged 6 to <72 Months) for Combined Seasons 2007/08 and 2008/09
Description: Virus-confirmed influenza illnesses were assessed and trivalent adjuvanted influenza vaccine (TIV-adj) was compared with Non-flu control vaccine and Flu-control vaccine for Influenza like illnesses for seasons 2007/08 and 2008/09.
Time Frame: 3 weeks after 2nd vaccination
Population: Analysis was done on Full Analysis Set
Measure: Number; unit: Number of subjects
Groups:
- TIV-adj (6 to < 36 Months): Subjects aged 6 to <36 months received 0.25 mL of each injection of Adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control (6 to < 36 Months): Subjects aged 6 to <36 months received 0.25 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- TIV-adj (6 to < 72 Months): Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Non-flu Control (6 to <72 Months): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
- Flu Control (6 to < 72 Months): Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
Arm/Group | TIV-adj (6 to < 36 Months) | Non-flu Control (6 to < 36 Months) | Flu-control (6 to < 36 Months) | TIV-adj (6 to < 72 Months) | Non-flu Control (6 to <72 Months) | Flu Control (6 to < 72 Months)
Number analyzed (Participants) | 1103 | 566 | 995 | 1937 | 993 | 1772
Number of subjects
  Subjects with ILI | 280 | 163 | 272 | 425 | 253 | 436
  Outpatient visits | 192 | 113 | 183 | 290 | 174 | 293
  Inpatient visits | 13 | 14 | 19 | 20 | 19 | 26
  Outcome (Recovered) | 269 | 159 | 267 | 414 | 248 | 431
  Outcome (Alive with sequelae) | 5 | 2 | 2 | 5 | 2 | 2
  Outcome (Lost to follow-up) | 3 | 0 | 1 | 3 | 0 | 1
  Outcome (ILI persisting) | 3 | 2 | 1 | 3 | 3 | 1
  Outcome (Not available) | 0 | 0 | 1 | 0 | 0 | 1

9. Secondary Outcome: Loss of Days of Usual Activity (Job, School, Day Care, Household/Family/Community Activities) Due to Influenza Like Illness (ILI) in Subjects in Aged 6 to <72 and 6 to <36 Months and in Direct Caregivers Living in the Household.
Description: as for outcome 8
Time Frame: 3 weeks after 2nd vaccination
Population: The analysis was done on Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TIV-adj | Non-flu Control | Flu-control
Number analyzed (Participants) | 425 | 253 | 436
Days
  Mean bed days (6 to <72 mths)(N=419,250,426) | 1.9 (2.3) | 2.3 (2.7) | 1.9 (2.4)
  Mean bed days (6 to <36 mths)(N=274,160,263) | 2.0 (2.5) | 2.1 (2.4) | 1.8 (2.4)
  Mean inactive days(6 to <72 mths)(N=417,249,427) | 3.1 (3.3) | 3.3 (3.5) | 2.9 (3.7)
  Mean inactive days(6 to <36 mths)(N=273,160,264) | 2.9 (3.3) | 3.0 (3.6) | 2.6 (3.3)

10. Secondary Outcome: Number of Events of Influenza Like Illness for Combined Seasons 2007/08 and 2008/09.
Description: The number of events of Influenza like Illness reported by subjects aged 6 to <72 months was assessed for combined seasons 2007/08 and 2008/09
Time Frame: 3 weeks after 2nd vaccination
Population: The analysis was done on Full Analysis Set
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | TIV-adj | Non-flu Control | Flu-control
Number analyzed (Participants) | 425 | 253 | 436
Events
  Mean ILI events (6 to <72 mths)(N=425,253,436) | 1.2 (0.5) | 1.3 (0.6) | 1.2 (0.5)
  Mean ILI events (6 to <36 mths)(N=280,163,272) | 1.3 (0.5) | 1.3 (0.6) | 1.3 (0.5)

11. Secondary Outcome: Immunogenicity of aTIV, Compared to Flu and Non-Flu-control, in Terms of GMRs, in Unprimed Subjects Aged 6 to <36 Months or Season 2008/09 (Homologous and Heterologous Strains)
Description: The immunogenicity was assessed in terms of Geometric mean titer ratios (GMRs) of study day 29/study day 1, study day 50/study day 1, study day 181/study day 1 were evaluated.
  The criteria for evaluation is GMR >2.5
Time Frame: On study days 1, 29, 50 and 181
Population: The analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Groups:
- TIV-adj: Subjects aged 6 to < 36 months received 0.25 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control: Subjects aged 6 to < 36 months received 0.25 mL of each injection of Non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-flu-control: Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 166 | 165 | 83
Ratios
  Day 29:1 A/Brisbane/2007 (A/H1N1) (N=165,163,82) | 17 [15 to 20] | 1.83 [1.57 to 2.13] | 1.03 [0.83 to 1.27]
  Day 50:1 A/Brisbane/2007 (A/H1N1) (N=160,162,78) | 83 [70 to 98] | 4.55 [3.84 to 5.39] | 1.11 [0.87 to 1.4]
  Day 181:1 A/Brisbane/2007 (A/H1N1) (N=161,163,80) | 19 [17 to 21] | 2.4 [2.11 to 2.73] | 1.02 [0.85 to 1.22]
  Day 29:1 A/Brisbane/2007 (A/H3N2) (N=165,163,82) | 15 [13 to 18] | 1.58 [1.38 to 1.81] | 1.07 [0.88 to 1.29]
  Day 50:1 A/Brisbane/2007 (A/H3N2) (N=160,162,78) | 86 [73 to 102] | 5.57 [4.73 to 6.55] | 1.04 [0.83 to 1.32]
  Day 181:1 A/Brisbane/2007 (A/H3N1) (N=161,163,80) | 30 [24 to 37] | 6.16 [4.97 to 7.63] | 2.1 [1.55 to 2.83]
  Day 29:1 B/Florida/2006 (N=165,163,82) | 2.11 [1.86 to 2.39] | 1.41 [1.24 to 1.6] | 1.06 [0.89 to 1.26]
  Day 50:1 B/Florida/2006 (N=160,162,78) | 14 [13 to 16] | 2.05 [1.81 to 2.31] | 1.02 [0.86 to 1.22]
  Day 181:1 B/Florida/2006 (N=161,163,80) | 4.22 [3.79 to 4.68] | 1.45 [1.31 to 1.61] | 1.05 [0.91 to 1.22]
  Day 29:1A/SolomonIsland/2006(A/H1N1)(N=165,163,82) | 2.1 [1.81 to 2.42] | 1.41 [1.22 to 1.62] | 0.97 [0.79 to 1.18]
  Day 50:1A/SolomonIsland/2006(A/H1N1)(N=160,162,78) | 18 [16 to 21] | 1.96 [1.7 to 2.25] | 0.98 [0.8 to 1.19]
  Day181:1A/SolomonIsland/2006(A/H1N1)(N=161,163,80) | 6.52 [5.79 to 7.34] | 1.6 [1.42 to 1.8] | 0.99 [0.84 to 1.16]
  Day 29:1 A/Wisconsin/2009 (A/H3N2)(N=165,163,82) | 4.56 [4.07 to 5.11] | 1.17 [1.05 to 1.31] | 0.95 [0.81 to 1.11]
  Day 50:1 A/Wisconsin/2009 (A/H3N2)(N=160,162,78) | 43 [37 to 50] | 3.01 [2.59 to 3.51] | 1.04 [0.84 to 1.29]
  Day181:1 A/Wisconsin/2009 (A/H3N2)(N=161,163,80) | 20 [16 to 25] | 5.06 [4.03 to 6.37] | 2.22 [1.61 to 3.06]
  Day 29:1 B/Brisbane/2008 (N=164,163,82) | 1.08 [1.04 to 1.11] | 1.02 [0.098 to 1.05] | 1 [0.96 to 1.05]
  Day 50:1 B/Brisbane/2008 (N=159,162,78) | 1.94 [1.8 to 2.08] | 1.11 [1.03 to 1.19] | 1.02 [0.93 to 1.14]
  Day181:1 B/Brisbane/2008 (N=160,163,80) | 1.04 [0.98 to 1.11] | 1.05 [0.98 to 1.11] | 1.26 [1.15 to 1.37]

12. Secondary Outcome: Immunogenicity of aTIV, Compared to Flu and Non-Flu-control, in Terms of Geometric Mean Titers (GMTs), in Unprimed Subjects Aged 6 to <36 Months for Season 2008/09 (Homologous and Heterologous Strains)
Description: Immunogenicity was analyzed in terms of Geometric Mean Titers (GMTs) as measured by hemagglutination inhibition (HI) assay. For each strain and each vaccine group, least squares GMTs, associated 2-sided 95% confidence interval were determined for all time points.
  Superiority analysis: GMT-TIV-adj/GMT-Flu-control >1 should be elicited to show that GMT-TIV-adj is superior to GMT-Flu-control
Time Frame: On study days 1, 29, 50 and 181
Population: The analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 166 | 165 | 83
Titers
  Day 1 A/Brisbane/2007 (A/H1N1) | 6.21 [5.33 to 7.24] | 7.52 [6.45 to 8.76] | 5.93 [4.8 to 7.33]
  Day 29 A/Brisbane/2007 (A/H1N1) (N=165,163,82) | 105 [82 to 136] | 14 [11 to 18] | 6.13 [4.33 to 8.69]
  Day 50 A/Brisbane/2007 (A/H1N1) (N=160,162,78) | 513 [405 to 652] | 35 [27 to 44] | 6.57 [4.71 to 9.16]
  Day 181 A/Brisbane/2007 (A/H1N1) (N=161,163,80) | 118 [95 to 146] | 18 [15 to 22] | 6.1 [4.51 to 8.25]
  Day 1 A/Brisbane/2007 (A/H3N2) | 5.85 [5.13 to 6.67] | 5.8 [5.09 to 6.6] | 5.66 [4.73 to 6.77]
  Day 29 A/Brisbane/2007 (A/H3N2) (N=165,163,82) | 90 [76 to 107] | 9.17 [7.71 to 11] | 6.04 [4.75 to 7.69]
  Day 50 A/Brisbane/2007 (A/H3N2) (N=160,162,78) | 510 [426 to 609] | 32 [27 to 39] | 6 [4.68 to 7.68]
  Day 181 A/Brisbane/2007 (A/H3N2) (N=161,163,80) | 176 [141 to 220] | 36 [29 to 45] | 12 [8.74 to 16]
  Day 1 B/Florida/2006 | 6.01 [5.59 to 6.45] | 6 [5.59 to 6.44] | 5.87 [5.32 to 6.47]
  Day 29 B/Florida/2006 (N=165,163,82) | 13 [11 to 15] | 8.45 [7.11 to 10] | 6.19 [4.87 to 7.87]
  Day 50 B/Florida/2006 (N=160,162,78) | 86 [74 to 100] | 12 [11 to 14] | 6.09 [4.95 to 7.49]
  Day 181 B/Florida/2006 (N=161,163,80) | 25 [22 to 29] | 8.72 [7.65 to 9.95] | 6.21 [5.16 to 7.48]
  Day 1 A/SolomonIslands/2006(A/H1N1) | 6.66 [5.56 to 7.98] | 8.19 [6.85 to 9.8] | 6.24 [4.87 to 8]
  Day 29 A/SolomonIslands/2006(A/H1N1)(N=165,163,82) | 14 [11 to 19] | 12 [8.69 to 15] | 6.08 [4.12 to 8.98]
  Day 50 A/SolomonIslands/2006(A/H1N1)(N=160,162,78) | 122 [94 to 157] | 16 [13 to 21] | 6.1 [4.27 to 8.73]
  Day181 A/SolomonIslands/2006(A/H1N1)(N=161,163,80) | 44 [34 to 55] | 13 [10 to 17] | 6.2 [4.46 to 8.61]
  Day 1 A/Wisconsin/2009 (A/H3N2) | 6.09 [5.26 to 7.06] | 6.74 [5.83 to 7.8] | 6.16 [5.03 to 7.53]
  Day 29 A/Wisconsin/2009 (A/H3N2)(N=165,163,82) | 28 [23 to 33] | 7.86 [6.57 to 9.39] | 5.87 [4.59 to 7.52]
  Day 50 A/Wisconsin/2009 (A/H3N2)(N=160,162,78) | 261 [218 to 313] | 20 [17 to 24] | 6.47 [5.03 to 8.32]
  Day181 A/Wisconsin/2009 (A/H3N2)(N=161,163,80) | 123 [97 to 156] | 34 [27 to 43] | 14 [9.81 to 19]
  Day 1 B/Brisbane/2008 (N=165,165,83) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Day 29 B/Brisbane/2008 (N=165,163,82) | 5.38 [5.21 to 5.56] | 5.08 [4.91 to 5.24] | 5 [4.78 to 5.23]
  Day 50 B/Brisbane/2008 (N=160,162,78) | 9.64 [8.96 to 10] | 5.55 [5.16 to 5.97] | 5.12 [4.63 to 5.68]
  Day181 B/Brisbane/2008 (N=161,163,80) | 5.21 [4.89 to 5.54] | 5.23 [4.92 to 5.56] | 6.28 [5.75 to 6.84]
Statistical Analysis 1: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H1N1)] = 0.83, 95% CI 2-sided [0.67 to 1.02]
Statistical Analysis 2: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H1N1)] = 7.63, 95% CI 2-sided [5.42 to 11]
Statistical Analysis 3: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H1N1)] = 15, 95% CI 2-sided [11 to 21]
Statistical Analysis 4: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H1N1)] = 6.48, 95% CI 2-sided [4.83 to 8.68]
Statistical Analysis 5: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H3N2)] = 1.01, 95% CI 2-sided [0.85 to 1.21]
Statistical Analysis 6: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H3N2)] = 9.82, 95% CI 2-sided [7.76 to 12]
Statistical Analysis 7: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H3N2)] = 16, 95% CI 2-sided [12 to 20]
Statistical Analysis 8: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Brisbane/2007 (A/H3N2)] = 4.92, 95% CI 2-sided [3.64 to 6.65]
Statistical Analysis 9: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[B/Florida/2006] = 1, 95% CI 2-sided [0.91 to 1.1]
Statistical Analysis 10: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[B/Florida/2006] = 1.5, 95% CI 2-sided [1.19 to 1.9]
Statistical Analysis 11: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[B/Florida/2006] = 6.99, 95% CI 2-sided [5.72 to 8.53]
Statistical Analysis 12: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[B/Florida/2006] = 2.92, 95% CI 2-sided [2.44 to 3.5]
Statistical Analysis 13: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1)] = 0.81, 95% CI 2-sided [0.64 to 1.04]
Statistical Analysis 14: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Solomon Islands/2006 (A/H1N1)] = 1.21, 95% CI 2-sided [0.83 to 1.78]
Statistical Analysis 15: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1] = 7.54, 95% CI 2-sided [5.33 to 11]
Statistical Analysis 16: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT[A/Solomon Islands/2006 (A/H1N1)] = 3.31, 95% CI 2-sided [2.4 to 4.55]
Statistical Analysis 17: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 0.9, 95% CI 2-sided [0.74 to 1.1]
Statistical Analysis 18: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; GMT; GMT[A/Wisconsin/2009 (A/H3N2)] = 3.54, 95% CI 2-sided [2.78 to 4.51]
Statistical Analysis 19: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 13, 95% CI 2-sided [10 to 16]
Statistical Analysis 20: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 3.6, 95% CI 2-sided [2.61 to 4.95]
Statistical Analysis 21: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1, 95% CI 2-sided [1 to 1]
Statistical Analysis 22: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1.06, 95% CI 2-sided [1.02 to 1.11]
Statistical Analysis 23: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1.74, 95% CI 2-sided [1.57 to 1.92]
Statistical Analysis 24: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <36 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1, 95% CI 2-sided [0.92 to 1.08]

13. Secondary Outcome: Percentage (95% CI) of Unprimed Subjects Aged 6 to <36 Months With HI Titer ≥1:40 in Season 2008/09 HI Assay(Homologous and Heterologous Strains)
Description: Percentage of subjects achieving seroprotection (i.e., with HI titer ≥1:40) at study day 1, study day 29, study day 50 and a study day 181 and associated 95% CI. The lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%.
Time Frame: On study days 1, 29, 50, 181
Population: The analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 166 | 165 | 83
Percentage of subjects
  Day 1 A/Brisbane/2007 (A/H1N1) | 5 [3 to 10] | 11 [7 to 17] | 5 [1 to 12]
  Day29 A/Brisbane/2007(A/H1N1)(N=165,163,82) | 92 [86 to 95] | 20 [14 to 27] | 6 [2 to 14]
  Day 50 A/Brisbane/2007 (A/H1N1) (N=160,162,78) | 100 [98 to 100] | 38 [31 to 46] | 6 [2 to 14]
  Day181A/Brisbane/2007(A/H1N1)(N=161,163,80) | 98 [94 to 99] | 25 [19 to 33] | 6 [2 to 14]
  Day1 A/Brisbane/2007(A/H3N2) | 4 [1 to 8] | 4 [1 to 8] | 2 [0 to 8]
  Day29 A/Brisbane/2007(A/H3N2)(N=165,163,82) | 95 [90 to 97] | 12 [7 to 18] | 4 [1 to 10]
  Day50 A/Brisbane/2007(A/H3N2)(N=160,162,78) | 99 [97 to 100] | 45 [37 to 53] | 4 [1 to 11]
  Day181A/Brisbane/2007(A/H3N2)(N=161,163,80) | 100 [98 to 100] | 45 [37 to 53] | 21 [13 to 32]
  Day 1 B/Florida/2006 | 2 [1 to 6] | 2 [0 to 5] | 1 [0.03 to 7]
  Day29 B/Florida/2006 (N=165,163,82) | 12 [8 to 18] | 12 [8 to 18] | 4 [1 to 10]
  Day50 B/Florida/2006 (N=160,162,78) | 88 [81 to 92] | 19 [13 to 25] | 3 [0 to 9]
  Day181B/Florida/2006 (N=161,163,80) | 40 [33 to 48] | 13 [9 to 20] | 3 [0 to 9]
  Day 1 A/SolomonIslands/2006(A/H1N1) | 5 [3 to 10] | 11 [7 to 17] | 5 [1 to 12]
  Day29A/Sol.Islands/2006(A/H1N1)(N=165,163,82) | 15 [10 to 21] | 13 [9 to 20] | 5 [1 to 12]
  Day50A/Sol.Islands/2006(A/H1N1) (N=160,162,78) | 95 [90 to 98] | 24 [18 to 31] | 5 [1 to 13]
  D181A/Sol.Islands/2006(A/H1N1) (N=161,163,80) | 61 [53 to 68] | 19 [13 to 26] | 5 [1 to 12]
  Day 1 A/Wisconsin/2009 (A/H3N2) | 4 [1 to 8] | 5 [2 to 9] | 2 [0 to 8]
  Day29 A/Wisconsin/2009(A/H3N2) (N=165,163,82) | 37 [30 to 45] | 6 [3 to 10] | 2 [0 to 9]
  Day50 A/Wisconsin/2009(A/H3N2) (N=160,162,78) | 100 [98 to 100] | 30 [23 to 37] | 4 [1 to 11]
  Day181A/Wisconsin/2009(A/H3N2) (N=161,163,80) | 99 [97 to 100] | 42 [34 to 50] | 23 [14 to 33]
  Day 1 B/Brisbane/2008 | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 4]
  Day29 B/Brisbane/2008 (N=165,163,82) | 1 [0.015 to 3] | 0 [0 to 2] | 0 [0 to 4]
  Day50 B/Brisbane/2008 (N=160,162,78) | 5 [2 to 10] | 0 [0 to 2] | 0 [0 to 5]
  Day181 B/Brisbane/2008 (N=161,163,80) | 0 [0 to 2] | 1 [0.016 to 3] | 6 [2 to 14]

14. Secondary Outcome: Percentage (95% CI) of Unprimed Subjects Aged 6 to <36 Months With Seroconversion From Baseline, for Season 2008/09 (Homologous and Heterologous Strains)
Description: HI assay was used for the analysis. Seroconversion is defined as negative pre-vaccination serum (<10)/ post-vaccination HI titer ≥1:40.
  Seroconversion is defined as either pre-vaccination HI titer <10 and a post-vaccination HI titer ≥1:40 or a prevaccination HI titer ≥10 and a minimum four-fold rise in post-vaccination HI antibody titer.
  The lower bound of the two-sided 95% confidence interval (CI) for the percentage of subjects achieving seroconversion for HI antibody should meet or exceed 40%.
Time Frame: On study days 1, 29, 50, 181
Population: The analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 165 | 163 | 82
Percentage of subjects
  Day29 A/Brisbane/2007(A/H1N1) | 92 [86 to 95] | 19 [13 to 26] | 1 [0.031 to 7]
  Day50 A/Brisbane/2007(A/H1N1)(N=160,162,78) | 100 [98 to 100] | 38 [30 to 46] | 1 [0.032 to 7]
  Day181A/Brisbane/2007(A/H1N1)(N=161,163,80) | 97 [93 to 99] | 24 [18 to 31] | 1 [0.032 to 7]
  Day29 A/Brisbane/2007(A/H3N2) | 93 [88 to 97] | 10 [6 to 16] | 1 [0.031 to 7]
  Day50 A/Brisbane/2007(A/H3N2)(N=160,162,78) | 98 [95 to 100] | 44 [36 to 52] | 1 [0.032 to 7]
  Day181A/Brisbane/2007(A/H3N2)(N=161,163,80) | 98 [94 to 99] | 42 [35 to 50] | 19 [11 to 29]
  Day29 B/Florida/2006 | 12 [8 to 18] | 12 [8 to 18] | 0 [0 to 4]
  Day50 B/Florida/2006 (N=160,162,78) | 88 [81 to 92] | 19 [13 to 25] | 0 [0 to 5]
  Day181B/Florida/2006 (N=161,163,80) | 39 [31 to 46] | 12 [7 to 18] | 1 [0.032 to 7]
  Day29A/Sol.Islands/2006(A/H1N1) | 14 [9 to 20] | 13 [8 to 19] | 0 [0 to 4]
  Day50A/Sol.Islands/2006(A/H1N1)(N=160,162,78) | 94 [89 to 97] | 23 [17 to 30] | 0 [0 to 5]
  Day181A/Sol.Islands/2006(A/H1N1)(N=161,163,80) | 60 [52 to 68] | 18 [12 to 25] | 0 [0 to 5]
  Day29 A/Wisconsin/2009(A/H3N2) | 36 [28 to 44] | 4 [1 to 8] | 0 [0 to 4]
  Day50 A/Wisconsin/2009(A/H3N2)(N=160,162,78) | 100 [98 to 100] | 27 [20 to 35] | 1 [0.032 to 7]
  Day181A/Wisconsin/2009(A/H3N2)(N=161,163,80) | 97 [93 to 99] | 39 [31 to 47] | 20 [12 to 30]
  Day29 B/Brisbane/2008 | 1 [0.015 to 3] | 0 [0 to 2] | 0 [0 to 4]
  Day 50:1 B/Brisbane/2008 (N=160,162,78) | 5 [2 to 12] | 0 [0 to 2] | 0 [0 to 5]
  Day181 B/Brisbane/2008 (N=161,163,80) | 0 [0 to 2] | 1 [0.016 to 3] | 6 [2 to 14]

15. Secondary Outcome: Immunogenicity of aTIV, Compared to Flu and Non-Flu-control, in Terms of GMTs, in Unprimed Subjects Aged 6 to <72 Months for Season 2008/09 (Homologous and Heterologous Strains)
Description: Immunogenicity was analyzed in terms of Geometric Mean Titers (GMTs) as measured by hemagglutination inhibition (HI) assay. For each strain and each vaccine group, least squares GMTs, associated 2-sided 95% confidence interval were determined for all time points Superiority analysis: GMT-TIV-adj/GMT-Flu-control >1 and GMT-TIV-adj/GMT-Non Flu-control >1 should be elicited to show that GMT-TIV-adj is superior to GMT-Flu-control/Non Flu-control.
Time Frame: On study days 1, 29, 50 , 181
Population: The analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 319 | 316 | 158
Titers
  Day 1 A/Brisbane/2007 (A/H1N1) | 9.63 [8.28 to 11] | 10 [8.59 to 12] | 9.48 [7.67 to 12]
  Day29A/Brisbane/2007(A/H1N1) (N=316,313,15 | 232 [185 to 291] | 36 [29 to 45] | 9.42 [6.85 to 13]
  Day50A/Brisbane/2007(A/H1N1) (N=310,309,150) | 735 [608 to 888] | 89 [74 to 108] | 9.91 [7.58 to 13]
  Day181A/Brisbane/2007(A/H1N1) (N=309,310,151) | 186 [155 to 225] | 43 [35 to 51] | 9.65 [7.41 to 13]
  Day1A/Brisbane/2007(A/H3N2) | 12 [10 to 15] | 12 [9.83 to 14] | 12 [8.98 to 15]
  Day 29 A/Brisbane/2007 (A/H3N2) (N=316,313,156) | 209 [167 to 261] | 33 [26 to 41] | 12 [8.83 to 17]
  Day 50 A/Brisbane/2007 (A/H3N2) (N=310,309,150) | 762 [634 to 915] | 95 [79 to 115] | 12 [9.18 to 15]
  Day 181 A/Brisbane/2007 (A/H3N2) (N=309,310,151) | 295 [245 to 356] | 94 [78 to 114] | 26 [20 to 34]
  Day 1 B/Florida/2006 | 6.37 [6.01 to 6.75] | 6.57 [6.2 to 6.96] | 6.41 [5.92 to 6.95]
  Day 29 B/Florida/2006 (N=316,313,156) | 21 [18 to 25] | 14 [12 to 16] | 6.54 [5.26 to 8.13]
  Day 50 B/Florida/2006 (N=310,309,150) | 109 [97 to 123] | 22 [19 to 25] | 6.67 [5.64 to 7.88]
  Day 181 B/Florida/2006 (N=309,310,151) | 32 [29 to 36] | 13 [11 to 14] | 6.92 [6.01 to 7.98]
  Day 1 A/SolomonIslands/2006(A/H1N1) | 11 [9.47 to 14] | 12 [9.89 to 14] | 10 [8.16 to 13]
  Day29 A/SolomonIslands/2006(A/H1N1)(N=316,313,150) | 40 [30 to 53] | 23 [18 to 31] | 10 [7.12 to 15]
  Day50 A/SolomonIslands/2006(A/H1N1)(N=310,309,150) | 228 [182 to 287] | 41 [33 to 51] | 11 [7.63 to 15]
  Day181A/SolomonIslands/2006(A/H1N1)(N=309,310,151) | 88 [70 to 109] | 28 [23 to 35] | 11 [7.76 to 14]
  Day 1 A/Wisconsin/2009 (A/H3N2) | 15 [12 to 18] | 15 [12 to 19] | 13 [9.97 to 18]
  Day 29 A/Wisconsin/2009 (A/H3N2) (N=316,313,156) | 98 [75 to 127] | 31 [24 to 40] | 13 [8.74 to 18]
  Day 50 A/Wisconsin/2009 (A/H3N2) (N=310,309,150) | 518 [420 to 639] | 70 [57 to 87] | 14 [10 to 19]
  Day181 A/Wisconsin/2009 (A/H3N2) (N=309,310,151) | 261 [212 to 322] | 98 [79 to 121] | 34 [26 to 46]
  Day 1 B/Brisbane/2008 | 5.05 [4.99 to 5.11] | 5.05 [5 to 5.11] | 5.08 [5 to 5.16]
  Day 29 B/Brisbane/2008 (N=316,313,156) | 6.31 [5.97 to 6.66] | 5.57 [5.28 to 5.89] | 5.11 [4.74 to 5.52]
  Day 50 B/Brisbane/2008 (N=310,309,150) | 12 [11 to 13] | 6.69 [6.23 to 7.17] | 5.2 [4.71 to 5.75]
  Day181 B/Brisbane/2008 (N=309,310,151) | 6.12 [5.77 to 6.49] | 5.67 [5.35 to 6.01] | 6.12 [5.64 to 6.65]
Statistical Analysis 1: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H1N1)] = 0.96, 95% CI 2-sided [0.78 to 1.19]
Statistical Analysis 2: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H1N1)] = 6.41, 95% CI 2-sided [4.69 to 8.76]
Statistical Analysis 3: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H1N1)] = 8.26, 95% CI 2-sided [6.36 to 11]
Statistical Analysis 4: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Brisbane/2007 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H1N1)] = 4.37, 95% CI 2-sided [3.38 to 5.65]
Statistical Analysis 5: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Brisbane/2007 (A/H3N2) in terms of Geometric Mean Titers GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H3N2)] = 1.05, 95% CI 2-sided [0.82 to 1.35]
Statistical Analysis 6: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H3N2)] = 6.42, 95% CI 2-sided [4.72 to 8.73]
Statistical Analysis 7: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H3N2)] = 7.98, 95% CI 2-sided [6.2 to 10]
Statistical Analysis 8: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Brisbane/2007 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Brisbane/2007 (A/H3N2)] = 3.13, 95% CI 2-sided [2.42 to 4.05]
Statistical Analysis 9: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Florida/2006] = 0.97, 95% CI 2-sided [0.9 to 1.05]
Statistical Analysis 10: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Florida/2006] = 1.56, 95% CI 2-sided [1.26 to 1.93]
Statistical Analysis 11: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Florida/2006] = 5, 95% CI 2-sided [4.25 to 5.88]
Statistical Analysis 12: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain B/Florida/2006 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Florida/2006] = 2.55, 95% CI 2-sided [2.22 to 2.93]
Statistical Analysis 13: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day1 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1)] = 0.96, 95% CI 2-sided [0.75 to 1.22]
Statistical Analysis 14: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1)] = 1.72, 95% CI 2-sided [1.17 to 2.51]
Statistical Analysis 15: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1)] = 5.58, 95% CI 2-sided [4.08 to 7.63]
Statistical Analysis 16: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Solomon Islands/2006 (A/H1N1) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Solomon Islands/2006 (A/H1N1)] = 3.11, 95% CI 2-sided [2.3 to 4.2]
Statistical Analysis 17: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 0.98, 95% CI 2-sided [0.74 to 1.3]
Statistical Analysis 18: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 3.14, 95% CI 2-sided [2.19 to 4.49]
Statistical Analysis 19: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 7.36, 95% CI 2-sided [5.51 to 9.82]
Statistical Analysis 20: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain A/Wisconsin/2009 (A/H3N2) in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [A/Wisconsin/2009 (A/H3N2)] = 2.66, 95% CI 2-sided [2 to 3.55]
Statistical Analysis 21: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 1 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 22: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 29 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1.13, 95% CI 2-sided [1.05 to 1.22]
Statistical Analysis 23: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 50 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1.79, 95% CI 2-sided [1.63 to 1.97]
Statistical Analysis 24: Comparison: TIV-adj vs Flu-control; To demonstrate superiority of immunogenicity of TIV-adj compared to Flu-control on Day 181 for strain B/Brisbane/2008 in terms of GMTs in subjects aged 6 to <72 months by HI assay; Test type: Superiority or Other; ANOVA; GMT [B/Brisbane/2008] = 1.08, 95% CI 2-sided [1 to 1.17]

16. Secondary Outcome: Immunogenicity of aTIV, Compared to Flu and Non-Flu-control, in Terms of GMRs, in Unprimed Subjects Aged 6 to <72 Months for Season 2008/09 (Homologous and Heterologous Strains)
Description: Hemagglutination Inhibition (HI) assay was used for the analysis. Geometric mean titer ratios (GMRs) of study day 29/study day 1, study day 50/study day 1, study day 181/study day 1 were evaluated.
  The criteria for evaluation is GMR >2.5
Time Frame: On study days 1, 29, 50, 181
Population: The analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 319 | 316 | 158
Ratios
  Day 29:1A/Brisbane/2007(A/H1N1;N=316,313,156) | 24 [21 to 27] | 3.6 [3.17 to 4.08] | 0.99 [0.83 to 1.18]
  Day 50:1A/Brisbane/2007(A/H1N1;N=10,309,150) | 76 [67 to 86] | 9 [7.89 to 10] | 1.02 [0.84 to 1.22]
  Day 181:1A/Brisbane/2007(A/H1N1;N=309,310,151) | 19 [17 to 21] | 4.31 [3.89 to 4.77] | 1.02 [0.88 to 1.17]
  Day 29:1A/Brisbane/2007(A/H3N2;N=316,313,156) | 17 [15 to 19] | 2.73 [2.4 to 3.09] | 1.03 [0.86 to 1.23]
  D50:1A/Brisbane/2007(A/H3N2;N=310,309,150) | 60 [52 to 69] | 8.03 [6.93 to 9.3] | 0.98 [0.8 to 1.21]
  Day 181:1A/Brisbane/2007(A/H3N2;N=309,310,151) | 24 [20 to 28] | 7.96 [6.71 to 9.44] | 2.21 [1.73 to 2.81]
  Day 29:1B/Florida/2006(N=316,313,156) | 3.32 [2.94 to 3.75] | 2.06 [1.83 to 2.33] | 1.03 [0.87 to 1.22]
  Day 50:1B/Florida/2006(N=310,309,150) | 17 [15 to 19] | 3.29 [2.98 to 3.63] | 1.03 [0.9 to 1.18]
  Day 181:1B/Florida/2006(N=309,310,151) | 5.05 [4.67 to 5.46] | 1.92 [1.78 to 2.08] | 1.06 [0.95 to 1.19]
  Day 29:1A/Sol.Island/2006(A/H1N1;N=316,313,156) | 3.51 [3.09 to 3.98] | 1.96 [1.72 to 2.22] | 0.99 [0.83 to 1.18]
  Day 50:1A/Sol.Island/2006A/H1N1;N=310,309,150) | 20 [18 to 22] | 3.49 [3.12 to 3.89] | 0.97 [0.83 to 1.14]
  Day 181:1A/Sol.Island/2006A/H1N1;N=309,310,151) | 7.63 [6.98 to 8.34] | 2.41 [2.2 to 2.63] | 1.01 [0.89 to 1.14]
  Day 29:1A/Wisconsin/2009(A/H3N2;N=316,313,156) | 6.59 [5.92 to 7.34] | 2.04 [1.83 to 2.27] | 0.93 [0.8 to 1.09]
  Day 50:1A/Wisconsin/2009(A/H3N2;N=310,309,150) | 34 [30 to 38] | 4.6 [4.07 to 5.2] | 0.98 [0.83 to 1.17]
  Day 181:1A/Wisconsin/2009(A/H3N2;N=309,310,151) | 18 [15 to 21] | 6.39 [5.36 to 7.6] | 2.59 [2 to 3.29]
  Day 29:1B/Brisbane/2008(N=315,313,156) | 1.25 [1.19 to 1.31] | 1.1 [1.05 to 1.16] | 1.01 [0.94 to 1.08]
  Day 50:1B/Brisbane/2008(N=309,309,150) | 2.38 [2.23 to 2.55] | 1.32 [1.24 to 1.42] | 1.02 [0.93 to 1.13]
  Day 181:1B/Brisbane/2008(N=308,310,151) | 1.21 [1.15 to 1.28] | 1.12 [1.06 to 1.19] | 1.21 [1.11 to 1.31]

17. Secondary Outcome: Percentages of Subjects With HI Titers ≥ 1:40 in Unprimed Subjects 6 to <72 Months of Age for Season 2008/09 Homologous and Heterologous Strains
Description: Hemagglutination Inhibition (HI) assay was used for the analysis.
  Percentage of subjects achieving seroprotection (i.e., with HI titer ≥1:40) at study day 1, study day 29, study day 50 and a study day 181 and associated 95% Confidence Intervals. The lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%.
Time Frame: On study days 1, 29, 50, 181
Population: The analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 319 | 316 | 158
Percentage of subjects
  Day1 A/Brisbane/2007(A/H1N1) | 20 [16 to 25] | 21 [17 to 26] | 16 [11 to 23]
  Day29A/Brisbane/2007(A/H1N1;N=316,313,156) | 96 [93 to 98] | 40 [35 to 46] | 17 [11 to 23]
  Day50A/Brisbane/2007(A/H1N1;N=310,309,150) | 100 [99 to 100] | 59 [54 to 65] | 17 [12 to 24]
  Day181A/Brisbane/2007(A/H1N1;N=309,310,151) | 98 [96 to 99] | 49 [43 to 54] | 18 [12 to 25]
  Day1A/Brisbane/2007(A/H3N2) | 23 [18 to 28] | 22 [17 to 27] | 20 [14 to 27]
  Day29A/Brisbane/2007(A/H3N2;N=316,313,156) | 96 [93 to 98] | 35 [30 to 40] | 21 [15 to 28]
  Day50A/Brisbane/2007(A/H3N2;N=310,309,150) | 99 [97 to 100] | 65 [60 to 71] | 21 [14 to 28]
  Day181A/Brisbane/2007(A/H3N2;N=309,310,151) | 100 [98 to 100] | 65 [60 to 70] | 41 [33 to 49]
  Day1B/Florida/2006 | 2 [1 to 4] | 2 [1 to 5] | 4 [1 to 8]
  Day29B/Florida/2006(N=316,313,156) | 28 [23 to 33] | 26 [21 to 31] | 4 [1 to 8]
  Day50B/Florida/2006(N=310,309,150) | 93 [89 to 95] | 38 [33 to 44] | 3 [1 to 8]
  Day181B/Florida/2006(N=309,310,151) | 52 [46 to 57] | 23 [18 to 28] | 4 [1 to 8]
  Day1A/Sol.Islands/2006(A/H1N1) | 21 [16 to 26] | 22 [17 to 27] | 18 [12 to 25]
  D29A/Sol.Islands/2006(A/H1N1;N=316,313,156) | 32 [27 to 38] | 24 [20 to 29] | 18 [12 to 25]
  D50A/Sol.islands/2006(A/H1N1;N=310,309,150) | 96 [94 to 98] | 45 [39 to 51] | 18 [12 to 25]
  D181A/Sol.Islands/2006(A/H1N1;N=309,310,151) | 72 [67 to 77] | 34 [29 to 40] | 18 [12 to 25]
  Day1A/Wisconsin/2009(A/H3N2) | 25 [21 to 31] | 25 [20 to 30] | 21 [15 to 28]
  Day29A/Wisconsin/2009(A/H3N2;N=316,313,156) | 60 [54 to 66] | 29 [24 to 34] | 21 [14 to 28]
  Day50A/Wisconsin/2009(A/H3N2;N=310,309,150) | 100 [98 to 100] | 54 [48 to 59] | 21 [15 to 29]
  D181A/Wisconsin/2009(A/H3N2;N=309,310,151) | 100 [98 to 100] | 63 [57 to 68] | 43 [35 to 51]
  Day1B/Brisbane/2008 | 0 [0 to 1] | 0 [0 to 1] | 1 [0.016 to 3]
  Day29B/Brisbane/2008(N=316,313,156) | 3 [2 to 6] | 1 [0 to 3] | 1 [0.016 to 4]
  Day50B/Brisbane/2008(N=310,309,150) | 10 [7 to 14] | 3 [1 to 5] | 0 [0 to 2]
  Day181B/Brisbane/2008(N=309,310,151) | 3 [1 to 5] | 3 [1 to 5] | 5 [2 to 10]

18. Secondary Outcome: Percentages of Subjects With Seroconversion and Vaccine Group Differences in Unprimed Subjects 6 to <72 Months of Age for Season 2008/09 (Homologous and Heterologous Strains)
Description: HI assay was used for the analysis. Seroconversion is defined as negative pre-vaccination serum (<10)/ post-vaccination HI titer ≥1:40.
  Seroconversion is defined as either pre-vaccination HI titer <10 and a post-vaccination HI titer ≥1:40 or a prevaccination HI titer ≥10 and a minimum 4-fold rise in post-vaccination HI antibody titer. The lower bound of the two-sided 95% confidence interval (CI) for the percentage of subjects achieving seroconversion for HI antibody should meet or exceed 40%.
Time Frame: On study days 1, 29, 50, 181
Population: The analysis was done on Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TIV-adj | Flu-control | Non-flu-control
Number analyzed (Participants) | 319 | 316 | 158
Percentage of subjects
  Day 29:1 A/Brisbane/2007 (A/H1N1; N=316,313,156) | 96 [93 to 98] | 40 [34 to 45] | 1 [0.016 to 4]
  Day 50:1 A/Brisbane/2007 (A/H1N1; N=310,309,150) | 100 [99 to 100] | 59 [53 to 64] | 1 [0 to 5]
  Day 181:1 A/Brisbane/2007 (A/H1N1; N=309,310,151) | 98 [96 to 99] | 48 [42 to 53] | 1 [0 to 5]
  Day 29:1 A/Brisbane/2007 (A/H3N2; N=316,313,156) | 94 [91 to 97] | 31 [26 to 37] | 1 [0.016 to 4]
  Day 50:1 A/Brisbane/2007 (A/H3N2; N=310,309,150) | 97 [95 to 99] | 63 [57 to 68] | 2 [0 to 6]
  Day 181:1 A/Brisbane/2007 (A/H3N2; N=309,310,151) | 93 [90 to 96] | 56 [51 to 62] | 23 [17 to 31]
  Day 29:1 B/Florida/2006 (N=316,313,156) | 28 [23 to 33] | 26 [21 to 31] | 0 [0 to 2]
  Day 50:1 B/Florida/2006 (N=310,309,150) | 93 [89 to 95] | 38 [32 to 43] | 1 [0.017 to 4]
  Day 181:1 B/Florida/2006 (N=309,310,151) | 50 [44 to 56] | 19 [15 to 24] | 1 [0 to 5]
  Day 29:1A/SolomonIsland/2006(A/H1N1;N=316,313,156) | 32 [27 to 37] | 24 [19 to 29] | 0 [0 to 2]
  Day 50:1A/SolomonIsland/2006(A/H1N1;N=310,309,150) | 96 [93 to 98] | 44 [39 to 50] | 0 [0 to 2]
  Day181:1A/SolomonIsland/2006(A/H1N1;N=309,310,151) | 72 [66 to 76] | 33 [27 to 38] | 0 [0 to 2]
  Day 29:1 A/Wisconsin/2009 (A/H3N2; N=316,313,156) | 58 [53 to 64] | 23 [19 to 28] | 1 [0.016 to 4]
  Day 50:1 A/Wisconsin/2009 (A/H3N2; N=310,309,150) | 98 [96 to 99] | 49 [43 to 54] | 2 [0 to 6]
  Day181:1 A/Wisconsin/2009 (A/H3N2;N=309,310,151) | 92 [89 to 95] | 52 [46 to 58] | 25 [18 to 33]
  Day 29:1 B/Brisbane/2008 (N=316,313,156) | 3 [2 to 6] | 1 [0 to 3] | 0 [0 to 2]
  Day 50:1 B/Brisbane/2008 (N=310,309,150) | 10 [7 to 14] | 3 [1 to 5] | 0 [0 to 2]
  Day181:1 B/Brisbane/2008 (N=309,310,151) | 2 [1 to 5] | 3 [1 to 5] | 5 [2 to 10]

19. Secondary Outcome: Number of Subjects With Local and Systemic Reactions for Egg and Cell Derived Inactivated Novel Swine Origin A/H1N1 Subunit Influenza Vaccines After Each Vaccination for All Seasons
Time Frame: 7 days post-vaccination
Population: Adequate data was not available to conduct this analysis.
Groups:
- Non-flu Control: Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of Novartis meningococcal C conjugate vaccine or tick-borne encephalitis vaccine
Arm/Group | TIV-adj | Flu-control | Non-flu Control
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Indirect Protective Effect of Fluad (NH Composition 2007/2008), Compared to Non-flu Control and Flu Control, in Connection to Household-contact Persons Via a Questioning of the Parents About ILI of Persons Living in the Same Household as the Study Child
Time Frame: 3 weeks after 2nd vaccination
Population: As per an amendment to the protocol, the Secondary efficacy endpoints were evaluated in enrolled subjects only and the household members were not included in the trial for the evaluation of indirect vaccine efficacy.
Arm/Group | TIV-adj | Non-flu Control | Flu-Control
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Incidence Rate of the 2009-2010 H1N1 Swine Pandemic Caused by a Novel Influenza A (H1N1) Virus of Swine Origin in Unprimed Children Aged 6 to <36 and 6 to <72 Months
Time Frame: 3 weeks after 2nd vaccination
Population: Adequate data was not available for assessing the incidence rates of the 2009-2010 swine pandemic caused by a novel influenza A (H1N1) virus of swine origin.
Groups:
- Flu-Control: Subjects aged 6 to < 36 months received 0.25 mL and those aged 36 to <72 months received 0.5 mL of each injection of
Arm/Group | TIV-adj | Non-flu Control | Flu-Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years (3 consecutive influenza seasons: 2007/08, 2008/09 and 2009/10).
Description: 15 subjects were excluded from safety analysis either because the subjects did not receive any of the study vaccines or the subjects received wrong vaccine at one of the visits.
Groups:
- TIV-adj_0.25: Subjects aged 6 to < 36 months received 0.25 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- TIV-adj_0.5: Subjects aged 36 to < 72 months received 0.5 mL of each injection of adjuvanted trivalent inactivated subunit influenza vaccine
- Flu-control_0.25: Subjects aged 6 to < 36 months received 0.25 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Flu-control_0.5: Subjects aged 36 to < 72 months received 0.5 mL of each injection of non-adjuvanted trivalent inactivated subunit influenza vaccine or non-adjuvanted trivalent inactivated split influenza vaccine
- Non-Flu-control (TBE/Men C Vaccine); Non-Flu-control (TBE Vaccine): Subjects aged 6 to <12 months received 2 doses of 0.5 mL of Novartis Meningococcal C conjugate vaccine and subjects aged 12 to <72 months received 2 doses of 0.25 mL of TBE vaccine
Arm/Group | TIV-adj_0.25 | TIV-adj_0.5 | Flu-control_0.25 | Flu-control_0.5 | Non-Flu-control (TBE/Men C Vaccine) | Non-Flu-control (TBE Vaccine)
Serious Adverse Events (participants affected / at risk) | 91/1177 | 31/835 | 104/1069 | 65/777 | 65/607 | 45/422
Other Adverse Events (participants affected / at risk) | 1101/1177 | 769/835 | 989/1069 | 686/777 | 567/607 | 375/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIV-adj_0.25 (N=1177) | TIV-adj_0.5 (N=835) | Flu-control_0.25 (N=1069) | Flu-control_0.5 (N=777) | Non-Flu-control (TBE/Men C Vaccine) (N=607) | Non-Flu-control (TBE Vaccine) (N=422)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 0
Developmental delay (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 2 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthropod infestation (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 8 | 3 | 7 | 0 | 3 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 3
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 14 | 1 | 13 | 3 | 8 | 2
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1 | 5 | 0 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hand-foot and mouth disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 12 | 8 | 39 | 40 | 33 | 31
Laryngitis (Infections and infestations) | 1 | 1 | 2 | 1 | 3 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pneumococcal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 5 | 3 | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pseudocroup (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 6 | 2 | 1 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Perineal Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Vaccination failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Paracentesis (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Acetonaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeding disorder of Infancy or Early childhood (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 0
Febrile convulsion (Nervous system disorders) | 2 | 1 | 4 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Attention deficit / Hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 2 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Child abuse (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0
Adenoidectomy (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0 | 0
Brain tumour operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Colonoscopy (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Exposure via ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Acquired epileptic aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIV-adj_0.25 (N=1177) | TIV-adj_0.5 (N=835) | Flu-control_0.25 (N=1069) | Flu-control_0.5 (N=777) | Non-Flu-control (TBE/Men C Vaccine) (N=607) | Non-Flu-control (TBE Vaccine) (N=422)
Conjunctivitis (Infections and infestations) | 164 | 83 | 156 | 65 | 91 | 45
Diarrhoea (Gastrointestinal disorders) | 309 | 45 | 260 | 35 | 147 | 10
Vomiting (Gastrointestinal disorders) | 188 | 64 | 166 | 70 | 102 | 23
Chills (General disorders) | 77 | 131 | 69 | 51 | 50 | 37
Fatigue (General disorders) | 1 | 338 | 2 | 224 | 2 | 122
Injection site erythema (General disorders) | 423 | 321 | 325 | 268 | 240 | 128
Injection site haemorrhage (General disorders) | 146 | 131 | 107 | 93 | 69 | 49
Injection site induration (General disorders) | 214 | 169 | 131 | 152 | 154 | 79
Injection site pain (General disorders) | 334 | 478 | 250 | 360 | 173 | 179
Injection site swelling (General disorders) | 123 | 156 | 90 | 128 | 83 | 54
Malaise (General disorders) | 0 | 196 | 1 | 120 | 0 | 64
Pyrexia (General disorders) | 482 | 299 | 412 | 183 | 221 | 125
Bronchitis (Infections and infestations) | 169 | 68 | 153 | 66 | 95 | 50
Ear infection (Infections and infestations) | 131 | 57 | 132 | 49 | 72 | 22
Gastroenteritis (Infections and infestations) | 178 | 75 | 152 | 85 | 94 | 36
Nasopharyngitis (Infections and infestations) | 153 | 78 | 161 | 74 | 89 | 36
Otitis media (Infections and infestations) | 250 | 109 | 226 | 110 | 130 | 62
Respiratory tract infection (Infections and infestations) | 76 | 29 | 62 | 37 | 44 | 17
Rhinitis (Infections and infestations) | 260 | 122 | 219 | 97 | 123 | 57
Tonsillitis (Infections and infestations) | 64 | 38 | 42 | 38 | 25 | 25
Upper respiratory tract infection (Infections and infestations) | 362 | 170 | 306 | 156 | 174 | 85
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 183 | 0 | 102 | 1 | 66
Crying (General disorders) | 373 | 5 | 325 | 3 | 163 | 0
Headache (Nervous system disorders) | 6 | 201 | 6 | 120 | 5 | 66
Somnolence (Nervous system disorders) | 381 | 1 | 315 | 1 | 186 | 0
Eating disorder (Psychiatric disorders) | 327 | 3 | 263 | 1 | 161 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 246 | 176 | 210 | 166 | 119 | 97
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 76 | 4 | 62 | 5 | 40 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 69 | 1 | 42 | 1 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 85 | 1 | 39 | 1 | 26
Viral infection (Infections and infestations) | 63 | 35 | 60 | 28 | 20 | 19
Enteritis (Gastrointestinal disorders) | 54 | 23 | 60 | 18 | 33 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days